CLINICAL TRIAL: NCT06535698
Title: A Single-Group Clinical Trial to Evaluate the Effect of an Oral Supplement to Provide Relief From Symptoms of Hormonal Imbalance.
Brief Title: Evaluating the Effect of a Supplement on Symptoms of Hormonal Imbalance.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Perelel Inc. (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20403
Record Dates: First submitted 2024-07-17; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Women's Health
Keywords: Hormonal Balance Support; Menstrual Cycle; Mood Swings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hormonal Balance Support Supplement (Experimental): Participants in this arm will receive Perelel Health hormonal balance support capsules. The dosage regimen is as follows:
  Week 1: 1 capsule daily in the evening Week 2: 2 capsules daily in the evening Weeks 3-12: 4 capsules daily (2 in the morning and 2 in the evening) The supplement contains Myo-inositol (1000 mcg), Metabolic balance blend (200 mcg) including Berberine HCl, Alpha lipoic acid, DIM (33'-Diindolylmethane), and D-chiro-inositol (25 mg). Other ingredients include Vegetable cellulose (capsule), plant cellulose, and L-leucine.
  Interventions: Dietary Supplement: Perelel Health Hormonal Balance Support

INTERVENTIONS:
Dietary Supplement: Perelel Health Hormonal Balance Support — The supplement contains Myo-inositol (1000 mcg), Metabolic balance blend (200 mcg) including Berberine HCl, Alpha lipoic acid, DIM (33'-Diindolylmethane), and D-chiro-inositol (25 mg). Other ingredients include Vegetable cellulose (capsule), plant cellulose, and L-leucine.

SUMMARY:
This is a virtual single-group trial lasting 12 weeks to evaluate the effects of Perelel Health's hormonal balance support on symptoms of hormonal imbalance and overall menstrual health.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported symptoms of hormonal imbalance (e.g., mood swings, irregular menstrual cycles)
* Generally healthy without uncontrolled chronic diseases
* Willing to avoid new hormonal balance treatments during the study
* Consistent use of current hormonal balance treatments for at least 3 months prior to the study

Exclusion Criteria:

* Chronic conditions preventing adherence to the protocol Diabetes
* Planned hormonal balance-related procedures during the study
* Started any new medications or supplements that target hormonal balance in the past 3 months
* Anyone with diabetes
* Severe allergies requiring EpiPen
* Pregnant, breastfeeding, or trying to conceive
* Recent surgeries or planned surgeries during the study
* Unwilling to follow the study protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Changes in Symptoms of Hormonal Imbalance | Baseline, Week 4, Week 8, Week 12
  Evaluation of the effect of Perelel Health hormonal balance support on symptoms of hormonal imbalance using a self-reported questionnaire.

SECONDARY OUTCOMES:
Changes in Overall Menstrual Health | Baseline, Week 4, Week 8, Week 12
  Assessment of the impact of Perelel Health hormonal balance support on menstrual health using a self-reported questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No